CLINICAL TRIAL: NCT05804110
Title: The Effect of Mindful Caring Education Program Based on Human Caring Theory on Nurses' Intentionality: An Action Research
Brief Title: The Effect of the Mindful Caring Education Program on Nurses' Intentionality
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma DURSUN ERGEZEN, Principal investigator, Akdeniz University
Other Study IDs: AkdenizF
Record Dates: First submitted 2023-03-23; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Nurses' Perceptions of Intentionality; the Facilitators of Intentionality; the Impediments to Intentionality; Effectiveness of Mindful Caring Education Program
Keywords: perceptions of intentionality; facilitators of intentionality; impediment to intentionality; mindful caring education program

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mindful Caring Education Program — A four-session education plan was prepared under the nature of action research. The Theory of Unitary Caring Science is transferred to practice through Caritas processes. In this context, ten Caritas processes and caring-healing modalities (meditation, reflection, etc.) were used in the study. The pilot study was carried out with six nurses face-to-face. The education program was conducted on an online platform. Each education took approximately 2.30-3 hours. The evaluation process in action research is an essential part of the change.

SUMMARY:
Intentionality is defined as the property of being about or directed toward a subject, as inherent in conscious states, beliefs, or creations of the mind. In nursing science, intentionality has been conceptualized as a dynamic and evolutionary antecedent of transpersonal caring in the mutual healing process. Intentionality is an ongoing process of discovering the nurse's self, purpose, and mission in life. The nurse's intentionality is a dynamic concept that evolves continuously. The nurse's cultural and ethnic background, philosophical and religious beliefs, life experiences, capacity for reflection, and self-awareness influence intentionality development and expression. It is recommended that nurses be encouraged to foster self-care and seek mentors and those who will support intentional care and healing practices. Also, breathing techniques, meditation, mindfulness, and self-reflection are recommended exercises for developing intentionality. Mindfulness is one way to cultivate personal knowing, awareness, and intentionality to facilitate growth and development in a transpersonal caring relationship. However, no research has been found to increase the nurse's mindful awareness or improve intentionality in the caring relationship. In this context, this research aimed to evaluate the effectiveness of mindful caring education on nurses' intentionality.

DETAILED DESCRIPTION:
Intentionality is defined as the property of being about or directed toward a subject, as inherent in conscious states, beliefs, or creations of the mind. In nursing science, intentionality has been conceptualized as a dynamic and evolutionary antecedent of transpersonal caring in the mutual healing process. Person experience stress, trauma, loss, and crisis in their lives in a caring relationship. These situations precipitate a need for healing. Intentionality enhances presence and brings a more profound strength and focus to each interaction. Authentic presence allows the nurse to hear the call. A nurse's goal and purposeful thought activate intentionality. The intentionality focuses on caring-healing consciousness. The nurse and person enter the caring moment. The nurse and the person enter a shared consciousness field.

Intentionality is an ongoing process of discovering the nurse's self, purpose, and mission in life. The nurse's intentionality is a dynamic concept that evolves continuously. The nurse's cultural and ethnic background, philosophical and religious beliefs, life experiences, capacity for reflection, and self-awareness influence intentionality development and expression. It is recommended that nurses be encouraged to foster self-care and seek mentors and those who will support intentional care and healing practices. Also, breathing techniques, meditation, mindfulness, and self-reflection are recommended exercises for developing intentionality. Mindfulness is one way to cultivate personal knowing, awareness, and intentionality to facilitate growth and development in a transpersonal caring relationship. Mindfulness is consistently paying attention to what is happening in the present moment. Mindfulness helps support full attention, deep understanding, and immediacy in caring practice. Practicing mindfulness, the nurse becomes fully available to see, understand, love, and care. Mindfulness facilitates attending to one's thoughts and actions in each moment to extend compassion to self, others, the world, and beyond.

Evidence shows that mindfulness-based interventions (MBI) help to reduce work-related stress, psychological distress, depression, burnout, and compassion fatigue. Also, MBI positively affects self-care awareness, emotion management, empathy satisfaction, professionals' receptivity, motivation, and responsiveness to others. However, no research has been found to increase the nurse's mindful awareness or improve intentionality in the caring relationship. The study aimed to explore nurses' perceptions of intentionality in caring relationships and the effectiveness of the mindful caring education program based on the Theory of Unitary Caring Science. In this context, the research questions are as follows:

Research Question 1. What are nurses' perceptions of intentionality in the caring relationship? Research Question 2. What are the facilitators of intentionality in the caring relationship? Research Question 3. What are the impediments to intentionality in the caring relationship? Research Question 4. Is a mindful caring education program effective in improving nurses' intentionality?

ELIGIBILITY:
Inclusion Criteria:

* At least 1 year of working experience in the clinic, willingness to participate in research.

Exclusion Criteria:

* The exclusion criteria were that the participants wanted to quit at any research stage and did not complete the education program.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nurses who care for adult patients in clinics.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
The perception of intentionality in the caring relationship | 3 month
  Since intentionality is a subjective phenomenon, one's feelings and thoughts should be analyzed with in-depth methods. For this purpose, individual interviews, observation, and vignettes were used as data collection methods. The questions in the data collection form to measure these variables are as follows:
  1. Semi-Structured Interview Questions Question 1. What does the concept of caring intentionality mean to you? Question 2. Do you have a caring story that has had a lasting impact on you? Could you share it with me?
  2. Field Notes:
     Encountered event/situation (place/time/person/dialogue/reactions):
     Observer's Comment:
  3. Vignettes
  Questions for vignettes are as follows:
  1. What did you think when you saw the patient?
  2. Can you describe how you felt when you saw the patient?
  3. What is the first situation/problem you want to solve when seeing the patient?
  4. What would you like to do for the patient's care?
The facilitators of intentionality in the caring relationship | 3 month
  Some factors facilitate intentionality in the caring relationship. These factors are seen in both the expressions and actions of the nurse. There is no objective measurement tool that can measure these factors. Therefore, this result is measured using semi-structured questions and field notes. The questions in the data collection form to measure these variables are as follows:
  1. Semi-Structured Interview Questions Question 1. Is there anything similar to your shared caring story facilitating your intentionality toward the patient? Could you share it with me?
  2. Field Notes
  Encountered event/situation (place/time/person/dialogue/reactions):
  Observer's Comment:
The impediments to intentionality in the caring relationship | 3 month
  Some factors hinder intentionality in the caring relationship. These factors are seen in both the expressions and actions of the nurse. There is no objective measurement tool that can measure these factors. Therefore, this result is measured using semi-structured questions and field notes. The questions in the data collection form to measure these variables are as follows:
  1. Semi-Structured Interview Questions Question: Is there anything similar to your shared caring story that hinders your intentionality toward the patient? Could you share it with me?
  2. Field Notes
  Encountered event/situation (place/time/person/dialogue/reactions):
  Observer's Comment:
Effectiveness of mindful caring education program | 3 month
  The effectiveness of the education program was evaluated using semi-structured interview questions, field notes, and vignettes. The same people filled out the same vignettes before and after the education sessions. The researchers criticized by comparing the responses given before and after the education program.
  1. Semi-Structured Interview Questions Question 1. What are your thoughts on a mindful caring education program?
  2. Field Notes
     Encountered event/situation (place/time/person/dialogue/reactions):
     Observer's Comment:
  3. Vignettes
  Questions for vignettes are as follows:
  1. What did you think when you saw the patient?
  2. Can you describe how you felt when you saw the patient?
  3. What is the first situation/problem you want to solve when seeing the patient?
  4. What would you like to do for the patient's care?

CONTACTS AND LOCATIONS:
Overall Officials: FATMA DURSUN ERGEZEN, phD, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aghebati N, Mohammadi E, Ahmadi F, Noaparast KB. Principle-based concept analysis: intentionality in holistic nursing theories. J Holist Nurs. 2015 Mar;33(1):68-83. doi: 10.1177/0898010114537402. Epub 2014 Jun 12. PMID 24923274
- [Result] Drick CA. Strengthening our awareness of presence through intentionality. Beginnings. 2014 Jun;34(3):22-4. No abstract available. PMID 25163192
- [Result] Dunn DJ. The intentionality of compassion energy. Holist Nurs Pract. 2009 Jul-Aug;23(4):222-9. doi: 10.1097/HNP.0b013e3181aecebb. PMID 19574759
- [Result] Watson J. Intentionality and caring-healing consciousness: a practice of transpersonal nursing. Holist Nurs Pract. 2002 Jul;16(4):12-9. doi: 10.1097/00004650-200207000-00005. PMID 12060941
- [Result] Zahourek RP. Intentionality in Healing--The Voices of Men in Nursing: A Grounded Theory Investigation. J Holist Nurs. 2015 Dec;33(4):308-23; quiz 324-5. doi: 10.1177/0898010115573665. Epub 2015 Mar 9. PMID 25755275
- [Result] Zahourek RP. Men in Nursing: Intention, Intentionality, Caring, and Healing: Emphasis on the Results of a Grounded Theory Study. Holist Nurs Pract. 2016 Sep-Oct;30(5):247-56. doi: 10.1097/HNP.0000000000000162. PMID 27501206
- [Result] Zahourek RP. Healing: through the lens of intentionality. Holist Nurs Pract. 2012 Jan-Feb;26(1):6-21. doi: 10.1097/HNP.0b013e31823bfe4c. PMID 22157505
- [Result] Zahourek RP. Theory: Intentionality the Matrix of Healing: A Theory Revised With Nonnurse Care Providers. J Holist Nurs. 2020 Sep;38(3):287-299. doi: 10.1177/0898010119892093. Epub 2019 Dec 9. PMID 31815573
- [Result] Deary L, Roche J, Plotkin K, Zahourek R. Intentionality and hatha yoga: an exploration of the theory of intentionality, the matrix of healing--a growth model. Holist Nurs Pract. 2011 Sep-Oct;25(5):246-53. doi: 10.1097/HNP.0b013e31822a02e0. PMID 21832929
- [Result] Zahourek RP. Intentionality: evolutionary development in healing: a grounded theory study for holistic nursing. J Holist Nurs. 2005 Mar;23(1):89-109. doi: 10.1177/0898010104272026. PMID 15665270